CLINICAL TRIAL: NCT04796246
Title: Leap Motion Controller on the Functionality Of Upper Limbs in Parkinson's Disease: A Randomized Clinical Trial
Brief Title: Leap Motion Controller on the Functionality of Upper Limbs in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fernanda Cechetti, Clinical Professor, Ph.D, Fernanda Cechetti, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24443019.7.0000.5345
Record Dates: First submitted 2020-07-21; First posted 2021-03-12 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease; Upper Extremity Dysfunction; Therapy-Related MDS
Keywords: Parkinson Disease; Upper Extremity Disfunction; Therapy-Related MDS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The proposed work will be characterized as a Randomized Clinical Trial, with evaluators outside the experimental groups (single-blind). The sample will be probabilistic, from individuals diagnosed with Parkinson's disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leap Motion Controller (Experimental): Intervention Group: which will receive treatment with Leap Motion Controller
  Interventions: Other: Leap Motion Controller; Other: Conventional Physiotherapy
- Conventional Physiotherapy (Active Comparator): Control Group: who will receive treatment with conventional physiotherapy.
  Interventions: Other: Leap Motion Controller; Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Leap Motion Controller — Training with the Leap Motion Controller instrument will be carried out first for 5 minutes, for a presentation and interaction of the virtual immersion with it, in the initial meeting. After the second meeting, the attendance protocol will be 16 sessions, this time being distributed as: first game lasting 7 minutes, second and third games lasting 6 minutes each and the last game lasting 8 minutes, totaling 27 minutes of intervention. Between games it was adopted about 2 minutes of rest.
Other: Conventional Physiotherapy — The conventional physiotherapy intervention will be based on the same activities developed (MMSS movements) of the IG: - First, attach pins with magnets with moving disc and after 1 minute and 25 seconds remove flower petals from inside a tube. The movements performed will be fine motricity, related to the tweezers handling (thumb and forefinger), alternating hands after 2 minutes and 30 minutes of play; - Hitting your hands on suddenly raised rulers, performing bilateral flexion / extension movements of the wrist simultaneously and alternating hands after 2 minutes and 30 minutes of play.

SUMMARY:
Is treatment with the Leap Motion Controller device effective for upper limb functionality in individuals with Parkinson's Disease?

The present study presents two hypotheses:

True hypothesis: There is an improvement in the functionality of MMSS after intervention with virtual reality? Null hypothesis: There is no improvement in the functionality of MMSS after intervention with virtual reality? The proposed work will be characterized as a Randomized Clinical Trial, with evaluators outside the experimental groups (single-blind). The sample will be probabilistic, from individuals diagnosed with Parkinson's disease.

DETAILED DESCRIPTION:
STUDY METHODOLOGY

1. RESEARCH DESIGN: The proposed work will be characterized as a Randomized Clinical Trial, with evaluators outside the experimental groups (single-blind). The sample will be probabilistic, from individuals diagnosed with Parkinson's disease.
2. TYPE OF STUDY: Randomized Clinical Trial.
3. AREA OF SCOPE: Major area: Health Sciences. Area: Physiotherapy and Occupational Therapy.
4. LOCATION: The place where the entire study will be carried out will be in the home environment of each research participant.
5. PARTICIPANTS: Participants will be recruited from an existing pre-existing list of research conducted on individuals with Parkinson's Disease from the UFCSPA. Individuals who: - are diagnosed with Parkinson's disease; - Classified as I-III on the Hoehn & Yahr motor staging scale; - Are over 18 years old (above this, without age restriction). - Residents in the city of Porto Alegre / RS. - Have signed the informed consent form (Appendix A). Individuals who: - Do not show the understanding of the games on the first day of familiarization; - Have a cerebral pacemaker implant; - Have recent injuries or limitations that make the MMSS impossible. - Do not perform / abstain from two appointments out of the 16 proposed in the intervention protocol, regardless of the group that will be allocated. The study will consist of two groups: intervention group (IG), which will receive treatment with Leap Motion Controller; and the control group (CG), who will receive treatment with conventional physiotherapy.
6. EVALUATION INSTRUMENTS: A participant identification form will be filled out, containing full name, date of birth, gender, address, telephone number, education, diagnosis, time of diagnosis, onset of symptoms (laterality), associated diseases, PD subtype and medicines. Individuals will be assessed for: the motor aspects of experiences and activities of daily living using the TEMPA test and the Unified Assessment Scale for Parkinson's Disease (MDS-UPDRS) part II; Motor Assessment and subtype of the disease, using the MDS-UPDRS scale III; motor staging of PD using the Hoehn & Yahr scale; muscle strength and endurance, using the handgrip dynamometer (TEMPA test); manual dexterity, through the Box and Block test and the Nine Hole Peg test; cognitive issues through the Montreal Cognitive Assessment (MoCA); and quality of life, through the Questionnaire on Parkinson's Disease (PDQ-39).
7. EXPECTED DURATION: The present research project contemplates different objectives, this being a study proposal to be developed during four years.
8. PROCEDURES: The formation of each of the groups will be done through the generation of a random sequence through the tool available at http://www.randomize.com. Therefore, individuals will be divided into two groups: Intervention Group and Control Group. Subsequently, the initial assessment will be made,TEMPA, MDS-UPDRS-II e III, motor staging of the disease (H&Y), Box and Block Test, Nine Hole Peg Test), MoCA and PDQ-39.The IG will carry out a 2-month intervention protocol, with 16 40-minute interventions, twice a week. The CG will perform a conventional physiotherapy protocol for the same period as the IG. Therefore, all groups will receive the same evaluation procedures that will be performed before the intervention (PRE), after the intervention (POST) and, finally, 30 days after the intervention (follow-up). The researchers responsible for the intervention will not be aware of the evaluations carried out and the evaluators will not be aware of the group to which the participant will belong. Both groups will be able to follow their routine activities (physical and / or physical therapy) and all procedures will be performed in the home environment of each research participant.
9. ETHICAL AND LEGAL PROCEDURES The study project in question will be submitted to the Research Ethics Committee of the Federal University of Health Sciences of Porto Alegre (UFCSPA) and will only be applied after due approval. All participants will be informed about the procedures, objectives, justifications, potential risks and benefits of their participation in the study. The research will not present risks to the participant, but if there is any discomfort during any activity, the treatment will be stopped immediately and the necessary measures taken. In addition, all participants must sign the informed consent form and receive a copy of it. The use of any type of image will not identify the participant and will only be used with written consent. The data in the medical record (name, telephone and address) will be used for screening in the identification and contact of individuals and stored in a database that will be accessed only by researchers.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnostic;
* Classified as I-III on the Hoehn & Yahr motor staging scale;
* Are over 18 years old (above this, without age restriction).
* Residents in the city of Porto Alegre / RS.
* Have signed an informed consent form.

Exclusion Criteria:

* Do not show the understanding of the games on the first day of familiarization;
* Have a cerebral pacemaker implant;
* Have recent injuries or limitations that make the MMSS impossible.
* Do not perform / abstain from two appointments out of the 16 proposed in the intervention protocol, regardless of the group that will be allocated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Test TEMPA (Test d'Évaluation des Membres Supérieurs de Personnes Agées) | Pre and Post Immediate intervention. 30 days after interventions.
  It is an instrument that serves to assess the degree of disability of the MMSS. It presents a manual on how to manage it, the necessary measures to make the box and where to dispose of each specific material of the tasks. The materials required for administering the test are as follows: 100 gram coffee pot, 1000 milliliter water jar, coffee spoon, cup, water glass, medicine bottle and 10 placebo capsules, white envelopes, seal, pencil , card game, coins (R $ 1, R $ 0.25, R $ 0.50, R $ 0.10), small glass jar (7 cm (cm) in diameter and 5 cm in height), small objects (toothpick, nut, safety pin, 2.5 cm diameter button and nail), piece of non-slip material and sheets for recording scores (MICHAELSEN et al., 2008). The test consists of performing bilateral and unilateral tasks, of the upper limbs.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Pre and Post Immediate intervention. 30 days after interventions.
  The updated MDS-UPDRS scale comprises four parts: Part I, the impact of non-motor aspects of daily life, part II, motor aspects of daily life, part III, motor assessment and part IV that corresponds to motor complications. However, only part II - motor aspects of daily life will be applied, which is designed to be a self-administered questionnaire, but can be reviewed by the researcher to ensure its clear and complete completion. And part III - motor evaluation, in which it has instructions for the evaluator to provide or demonstrate to the individual and is completed by the evaluator. A higher score corresponds to a corresponding worse state.

OTHER OUTCOMES:
Hoehn & Yahr Scale | Pre and Post Immediate intervention. 30 days after interventions.
  The Hoehn & Yahr (H&Y) staging scale serves to classify and determine which motor stage of Parkinson's disease the individual is in. It is an easy and quick scale to be applied, which has its modified form, comprising five stages of classification to assess the severity of PD, and is based mainly on the signs and symptoms to assess the individual's level of disability. Individuals rated on the scale between one and three are in stages of mild to moderate disability, while those with stages four and five fall into severe disability.
Box and Block Test | Pre and Post Immediate intervention. 30 days after interventions.
  For the application of the manual dexterity test, a wooden box with a length of 53.7 cm is required, with a partition also made of wood higher than the edges of the box, separating it into two compartments of equal dimensions. The blocks also made of wood and in the form of colored cubes (primary colors) of 2.5 cm on a side are 150 in number, divided equally by color. As a prerequisite for the application of the test, a quiet environment is necessary, with the subject being seated in a chair suitable for his / her height. The box must be placed horizontally in front of him so that he has a full view of the area and equipment in question.
Nine Hole Peg Test | Pre and Post Immediate intervention. 30 days after interventions.
  The test that assesses manual dexterity consists of nine pins and a plate with nine holes, in which the individual is instructed to take one pin at a time and insert it into the holes contained in the plate and then, later remove the pins and return it. them to the place of origin. The execution time is timed by the researcher.
Montreal Cognitive Assessement - MoCA | Pre and Post Immediate intervention. 30 days after interventions.
  The MoCA measures eight cognitive domains, which are scored within a range of 0 to 30 points (higher scores indicating better function): short-term memory (delayed recall, 5 points); visuospatial skills (cube design, 1 point, clock design, 3 points); executive function (trail test, 1 point; phonemic verbal fluency, 1 point; verbal abstraction, 2 points); attention, concentration and working memory (cancellation, 1 point; subtraction, 3 points; digit range, 2 points); language (nomination, 3 points; sentence repetition, 2 points); and orientation in time (3 points) and space (3 points).
Parkinson's Disease Questionnaire - PDQ-39 | Pre and Post Immediate intervention. 30 days after interventions.
  The Parkinson's Disease questionnaire, PDQ-39, consists of 39 questions covering the topics: mobility, activities of daily living, emotional well-being, social support, body discomfort, stigma, cognition and communication. The individual identifies how often in the last month he found himself in the situations mentioned. The options are never (0 points), rarely (1 point), sometimes (2 points), often (3 points) and always (4 points). Between 0 and 100 the lowest score corresponds to the highest quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Philipe Souza Correa, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided